CLINICAL TRIAL: NCT03614793
Title: A Prospective Trial of Cooled Radiofrequency Ablation of Medial Branch Nerves Versus Facet Joint Injection of Corticosteroid for the Treatment of Lumbar Facet Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Zack McCormick, Associate Professor, Spine and Pain Medicine Director, Clinical Spine Research Director, Interventional Spine and Musculoskeletal Medicine Fellowship, Division of Physical Medicine and Rehabilitation University of Utah School of Medicine, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111315
Record Dates: First submitted 2018-07-12; First posted 2018-08-03 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lumbar Facet Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooled Radiofrequency Ablation Procedure (Active Comparator): Cooled Radiofrequency Ablation (C-RFA) Procedure:
  This is performed under image (x-ray) guidance for the accuracy of needle placement. A Cooled Radiofrequency electrode will be placed at the surface of the facet joint. After appropriate electrode positioning, a local anesthetic (lidocaine) will be injected through the needle to take away pain during the ablation. Once the procedure is completed, all needles will be removed and additional local anesthetic (bupivacaine) will be injected. No corticosteroids will be injected.
  Interventions: Procedure: Cooled Radiofrequency Ablation of Medial Branch Nerves versus Facet Joint Injection of Corticosteroid for the Treatment of Lumbar Facet Syndrome
- Facet Joint Inject Procedure (Active Comparator): Facet joint injection (FJI) Procedure:
  This is performed under image guidance (x-ray) for the accuracy of needle placement. A needle will be carefully placed in the facet joint(s) causing pain. Contrast will be injected to confirm the ideal needle placement. The injection will then be completed with triamcinolone (steroid) and lidocaine. This technique will be repeated for each facet joint injected. For bilateral low back pain, a maximum of 4 facet joints (two on each side) will be treated. For unilateral low back pain, up to 3 facet joints will be treated.
  Interventions: Procedure: Cooled Radiofrequency Ablation of Medial Branch Nerves versus Facet Joint Injection of Corticosteroid for the Treatment of Lumbar Facet Syndrome

INTERVENTIONS:
Procedure: Cooled Radiofrequency Ablation of Medial Branch Nerves versus Facet Joint Injection of Corticosteroid for the Treatment of Lumbar Facet Syndrome — Radio frequency ablation (RFA) is a medical procedure in which heat is generated from high frequency electrical current in order to lesion (burn) nervous tissue.

SUMMARY:
Chronic, non-neurogenic low back pain (CLBP) is a common condition that affects many individuals across their lives. The lumbar facet joint has been implicated as an important source of CLBP, with a prevalence of 15-45%. Elements of clinical history, physical examination, and imaging (radiographs, standard CT scan, standard MRI sequences) provide poor diagnostic specificity for pain of lumbar zygapophysial joint (Z-joint) origin. Thus, clinicians have traditionally relied upon MBN blocks to confirm or refute this diagnosis. The reference standard for the diagnosis of lumbar Z-joint pain is a positive response to dual comparative MBN blocks, which requires pain reduction of great than or equal to 80% of concordant duration to that expected of two different local anesthetics on independent occasions. Further, dual comparative MBN blocks have a high positive predictive value for determining the clinical outcome of lumbar MBN RFA for the treatment of lumbar Z-joint pain; when patients are appropriately selected using this reference standard and rigorous MBN RFA technique is implemented according to practice guidelines, studies demonstrate excellent clinical outcomes.

DETAILED DESCRIPTION:
Chronic, non-neurogenic low back pain (CLBP) is a common condition that affects many individuals across their lives. The lumbar facet joint has been implicated as an important source of CLBP, with a prevalence of 15-45%. Elements of clinical history, physical examination, and imaging (radiographs, standard CT scan, standard MRI sequences) provide poor diagnostic specificity for pain of lumbar zygapophysial joint (Z-joint) origin. Thus, clinicians have traditionally relied upon MBN blocks to confirm or refute this diagnosis. The reference standard for the diagnosis of lumbar Z-joint pain is a positive response to dual comparative MBN blocks, which requires pain reduction of great than or equal to 80% of concordant duration to that expected of two different local anesthetics on independent occasions. Further, dual comparative MBN blocks have a high positive predictive value for determining the clinical outcome of lumbar MBN RFA for the treatment of lumbar Z-joint pain; when patients are appropriately selected using this reference standard and rigorous MBN RFA technique is implemented according to practice guidelines, studies demonstrate excellent clinical outcomes.

In additional to MBN RFA, lumbar facet joint injection of corticosteroid is another commonly used treatment strategy for lumbar facet joint pain related to osteoarthritis. While clinical outcome studies of facet joint injection with corticosteroid have generally shown only modest outcome improvements, this literature is generally flawed by invalid selection protocols that do not require dual comparative MBN blocks in order to confirm the diagnosis of pain specific to the lumbar facet joint(s).

Despite the widespread use of these two techniques (lumbar MBN RFA vs. facet joint corticosteroid injection), the two techniques have never been compared in an appropriately-designed head-to-head study. The sole outcome study comparing these two treatment methods used an invalid selection protocol of one positive MBN block, requiring only 50% relief in pain and not of concordant duration with that expected by the local anesthetic used; in addition, a single RFA lesion was applied with a 20g conventional RFA electrode and fluoroscopic images were not published, so it is unclear if parallel electrode technique was used, as is necessary with conventional RFA. This invalid patient selection and RFA technique protocol is similar to that used in the Mint Trials, which has led to a broad call for improving such standards in research and clinical care by a multitude of experts representing interventional pain, spine, and radiology specialty societies. As such, an appropriately designed head-to-head trial in warranted.

Furthermore, while the conventional RFA modality has been studied extensively for MBN RFA, minimal outcome literature on the effectiveness of C-RFA technology has been published. C-RFA is similar in mechanism to conventional RFA: a thermal lesion is created by applying radiofrequency energy through an electrode placed at a target structure. In C-RFA, a constant flow of ambient water is circulated through the electrode via a peristaltic pump, maintaining a lowered tissue temperature by creating a heat sink. By removing heat from tissues immediately adjacent to the electrode tip, a lower lesioning temperature is maintained, resulting in less tissue charring adjacent to the electrode, less tissue impedance and more efficient heating of target tissue. The volume of tissue heated, and the resultant thermal lesion size is substantially larger with C-RFA, conferring an advantage over conventional RFA. Further, given the spherical geometry and forward projection the C-RFA lesions beyond the distal end of the electrode, the RFA probe can be positioned at a range of possible angles and still capture the target neural structure, whereas more fastidious, parallel positioning is required with conventional RFA. These technical advantages increase the probability of successful denervation of neural pain generators that have variability in anatomic location, as is the case with facet syndromes in which significant osteoarthritis is present, which is associated with joint hypertrophy and osteophyte formation. Additionally, a longer lesion of the MBN may be more reliably achieved with C-RFA compared to conventional RFA, potentially resulted in greater treatment durability, as the recurrent of facetogenic pain after successful denervation is related to reinnervation by nerve re-growth to bridge the gap created by the lesion. Consistent with this technical advantage, there is preliminary evidence for superiority of C-RFA compared to both conventional RFA and other novel RFA techniques in the treatment of sacroiliac joint-mediated pain.

Lumbar facet joint pain is a common and costly cause of chronic low back pain. Lumbar MBN RFA and facet joint injection of steroid are two commonly used treatment strategies for lumbar facet-mediated pain, yet the two techniques have never been compared in an appropriately-designed head-to-head trial. Further there is minimal clinical outcome literature describing the effectiveness of MBN C-RFA despite its technical advantages over conventional MBN RFA. We will determine if individuals with lumbar facet syndrome who are treated with MBN C-RFA compared to face joint injection of corticosteroid have a greater likelihood of experiencing meaningful relief of low back pain symptoms, functional improvement, and reduction of analgesic medication use at both short and long-term follow-up. Answering this clinical question will help determine which standard of care technique is superior, such that patients with lumbar facet syndrome can get be offered the best treatment available.

As such, the goal of the proposed study is to determine if individuals with lumbar facet syndrome who are treated with C-RFA of the MBNs compared to face joint injection of corticosteroid have a greater likelihood of experiencing meaningful relief of low back pain symptoms, functional improvement, and reduction of analgesic medication use at both short and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged > 21 capable of understanding and providing consent in English and capable of complying with the outcome instruments used.
* Axial (non-radicular) back pain for at least 3 months (ie Chronic Low Back Pain), with pain lasting at least half of the days within those 3 months, that did not respond to conventional treatment such as physical therapy, oral analgesic agents, and non-invasive adjunctive treatments. The pain can be unilateral or bilateral. The pain can also include referred lower limb pain.
* 7-day worst numeric pain rating score (NPRS) for back pain of 5/10 or greater at baseline evaluation.
* Positive responses to dual comparative diagnostic MBN blocks using 0.5mL of 0.5% bupivacaine and 4% lidocaine, on respective encounters on separate days, at each of the appropriate MBNs. The blocks are administered in a double-blind fashion so that neither the subject nor the independent assessor is aware of the local anesthetic used.

Exclusion Criteria:

* Focal neurologic signs or symptoms.
* Radiologic evidence of a symptomatic herniated disc or nerve root impingement related to spinal stenosis.
* Active systemic or local infections at the site of proposed needle and electrode placement.
* Coagulopathy or other bleeding disorder.
* Receipt of remuneration for their pain treatment (e.g. disability, worker's compensation, auto injury in litigation or pending litigation).
* History of any lumbar or lower thoracic fusion surgery or placement of other hardware.
* > Grade 2 Spondylolisthesis at an affected or adjacent level.
* Cobb angle >10 degrees.
* Sagittal vertical axis angle >5 degrees
* BMI >40.
* Incarceration.
* Cognitive deficit affecting ability to complete the assessment instruments.
* Inability to read English and complete the assessment instruments.
* Allergy to local anesthetics.
* Chronic widespread pain or somatoform disorder (e.g. fibromyalgia).
* Prior lumbar MBN radiofrequency neurotomy.
* Addictive behavior, severe clinical depression, anxiety, or any mental health condition with psychotic features.
* Possible pregnancy or other reason that precludes the use of fluoroscopy.
* Daily chronic opiate use of >50 morphine equivalents.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] McCormick ZL, Conger A, Kendall R, Wagner G, Henrie AM, Littell M, Sperry BP, Petersen R, Cooper AN, Teramoto M, Burnham TR. A pragmatic randomized prospective trial of cooled radiofrequency ablation of the medial branch nerves versus facet joint injection of corticosteroid for the treatment of lumbar facet syndrome: 12 month outcomes. Pain Med. 2023 Dec 1;24(12):1318-1331. doi: 10.1093/pm/pnad107. PMID 37578437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started in October of 2018. Out of 1128 participants, 1089 did not meet eligibility criteria and 35 weren't interested. 39 were randomized. 6 withdrew from the FJI group before treatment, 5 due to insurance denial of FJI (started during the study recruitment period) and 1 who lost interest in the study.
  Of the 13 remaining patients in the FJI group, 1 individual was lost to follow-up after receiving FJI treatment. Consequently, a total of 32 patients were analyzed in this study.
Pre-assignment Details: During screening, some participants were discontinued before randomization. The most common reasons were:
  Insurance denied payment of second medial branch block, Participant had a Cobb angle greater than 10, Participant had concurrent radiculopathy, Negative medial branch block, Did not meet eligibility criteria
Groups:
- Cooled Radiofrequency Ablation Procedure: Cooled Radiofrequency Ablation (C-RFA) Procedure:
  This is performed under image (x-ray) guidance for the accuracy of needle placement. A Cooled Radiofrequency electrode will be placed at the surface of the facet joint. After appropriate electrode positioning, a local anesthetic (lidocaine) will be injected through the needle to take away pain during the ablation. Radiofrequency ablation (RFA) is a medical procedure in which heat is generated from high-frequency electrical current to lesion (burn) a targeted nerve. Once the procedure is completed, all needles will be removed and additional local anesthetic (bupivacaine) will be injected. No corticosteroids will be injected.
Period: Overall Study
Arm/Group | Cooled Radiofrequency Ablation Procedure | Facet Joint Inject Procedure
Started | 20 | 19
Completed | 19 | 6
Not Completed | 1 | 13
Not completed — Lost to Follow-up | 1 | 2
Not completed — Lack of Efficacy | 0 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Insurance denied coverage of the procedure | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Cooled Radiofrequency Ablation Procedure: Cooled Radiofrequency Ablation (C-RFA) Procedure:
  Radiofrequency ablation (RFA) is a medical procedure in which heat is generated from high-frequency electrical current to lesion (burn) a targeted nerve.
  The procedure was performed under fluoroscopy guidance for the accuracy of needle placement. A Cooled Radiofrequency electrode was placed at the surface of the facet joint. After appropriate electrode positioning, a local anesthetic (lidocaine) was injected through the needle to help with pain during the ablation. Once the procedure was completed, all needles were removed and additional local anesthetic (bupivacaine) was injected. No corticosteroids were injected.
- Facet Joint Inject Procedure: Facet joint injection (FJI) Procedure:
  The procedure was performed under fluoroscopy guidance for the accuracy of needle placement. A needle was carefully placed in the facet joint(s) causing pain. Contrast dye was injected to confirm the ideal needle placement. The injection was then completed with triamcinolone (steroid) and lidocaine. This technique was repeated for each facet joint injected. For bilateral low back pain, a maximum of 4 facet joints (two on each side) were treated. For unilateral low back pain, up to 3 facet joints were treated.
- Total: Total of all reporting groups
Arm/Group | Cooled Radiofrequency Ablation Procedure | Facet Joint Inject Procedure | Total
Number analyzed (Participants) | 20 | 12 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (12.4) | 62.4 (14.6) | 62.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 4 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 12 | 32
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.7 (5.3) | 25.7 (5.3) | 27.2 (5.3)
Duration of low back pain [Mean (Standard Deviation); unit: years] | 4.9 (1.1) | 5.4 (0.9) | 5.2 (1)
Laterality of pain [Number; unit: Number of participants]
  Unilateral | 10 | 3 | 13
  Bilateral | 10 | 9 | 19
Number of painful facet joints [Mean (Standard Deviation); unit: Number of painful facet joints] | 2.1 (0.3) | 1.9 (0.3) | 2 (0.3)
Opioid use [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 3
  No | 19 | 10 | 29
Back Pain NPRS 7-Day Average [Mean (Standard Deviation); unit: Pain Scale 0 to 10] — This is a scale from 0 to 10, with 0 being no back pain at all and 10 being the worst back pain imaginable. The participant is asked to provide the average of their back pain over the previous 7 days.
  Pain Scale 0 to 10 | 4.9 (1.4) | 6.2 (2.2) | 5.6 (1.8)
Oswestry Disability Index Score [Mean (Standard Deviation); unit: units on a scale] | 15.1 (5.0) | 19.5 (8.6) | 17.3 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: This is a scale from 0 to 10, with 0 being no back pain at all and 10 being the worst back pain imaginable
  The primary outcome for this study was the proportion of participants within each group (C-RFA and FJI) who experienced a greater than or equal to 50% reduction in NPRS score at 3 months. Participants were asked to rate their pain over the past 7 days on a scale from 0 to 10.
Time Frame: 3 Months
Population: Out of 1128 patients assessed for eligibility, 1089 were not eligible. 39 randomized: 20 to C-RFA and 19 to FJI. 6 withdrew from the FJI group: 5 due to insurance denial and 1 opted out. Of the 13 remaining patients in the FJI group, 1 was lost to follow-up after treatment. A total of 32 patients were analyzed in this study: 20 C-RFA and 12 FJI. Due to the insurance coverage change for FJI, 1:1 randomization was no longer possible. Enrollment ended early.
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency Ablation Procedure | Facet Joint Inject Procedure
Number analyzed (Participants) | 20 | 12
Participants | 14 | 3

2. Secondary Outcome: Decrease in Oswestry Disability Index (ODI) Score
Description: ODI Percentage 0% to 20%: minimal disability: The patient can cope with most living activities. Usually, no treatment is indicated apart from advice on lifting sitting and exercise.
  21%-40%: moderate disability: The patient has more pain and difficulty with sitting, lifting and standing. Travel and social life are more difficult and they may be disabled from work. Personal care, sexual activity and sleeping are not grossly affected and the patient can usually be managed by conservative means.
  41%-60%: severe disability: Pain remains the main problem in this group but activities of daily living are affected. These patients require a detailed investigation.
  61%-80%: crippled: Back pain impinges on all aspects of the patient's life. Positive intervention is required.
  81%-100%: These patients are either bed-bound or exaggerating their symptoms.
  This secondary outcome measured how many participants had an equal to or greater than 30% decrease in their ODI score.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency Ablation Procedure | Facet Joint Inject Procedure
Number analyzed (Participants) | 20 | 12
Participants | 3 | 8

3. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC questionnaire allows participants to give their opinion on how well the treatment worked for them. Participants are asked to rate the status of their lower back pain after treatment: Very much worse, Much worse, Minimally worse, No change, Minimally improved, Much improved and Very much improved.
  The variable for this outcome was how many participants reported equal to or greater than a 6, which would be "Much improved" or "Very much improved."
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency Ablation Procedure | Facet Joint Inject Procedure
Number analyzed (Participants) | 20 | 12
Participants | 11 | 4

4. Secondary Outcome: Numeric Pain Rating Scale (NPRS) Point Change
Description: This outcome was measured at 6 months from the NPRS scale, 0 being no pain to 10 being the worst pain imaginable, to see how many participants had an equal to or greater than a 2-point reduction in their pain compared to baseline.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency Ablation Procedure | Facet Joint Inject Procedure
Number analyzed (Participants) | 20 | 12
Participants | 13 | 3

5. Secondary Outcome: Global Impression of Change (PGIC)
Description: PGIC survey-based assessment of subjective improvement in overall symptoms. This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status.
Time Frame: 2 year
Reporting Status: Not Posted

6. Secondary Outcome: Adverse Events
Description: Report immediate, short-term, and long-term adverse effects, using a standardized survey that includes a comprehensive query of known adverse events associated with systemic steroid effects
Time Frame: 2 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 Months
Description: As this was a pragmatic comparative trial of standard-of-care procedures, only specific Adverse Events were to be recorded: spinal infection, epidural hematoma, and neurological damages to the spinal nerve root(s) at the treated level(s).
Arm/Group | Cooled Radiofrequency Ablation Procedure | Facet Joint Inject Procedure
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03614793/Prot_SAP_001.pdf